CLINICAL TRIAL: NCT03794050
Title: Effects of Age, Fitness Level, and Modality on Physiological Response to Acute Exercise
Brief Title: Comparing Acute Aerobic and Resistance Exercise
Acronym: CAARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to SARS-CoV-2 pandemic research restrictions placed by university, we were unable to complete enrollment of all participants in a timely manner. Data analyses and publications will occur with the participants who did complete the study.
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Melissa M Markofski, Assistant Professor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001191
Record Dates: First submitted 2018-12-17; First posted 2019-01-04 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Exercise Physiology
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistance training exercise (Experimental): All participants complete one session of resistance training exercise
  Interventions: Other: Resistance training exercise
- aerobic training exercise (Experimental): All participants complete one session of aerobic training exercise
  Interventions: Other: Aerobic training exercise

INTERVENTIONS:
Other: Resistance training exercise — randomized complete crossover for acute resistance training exercise session
  Arms: resistance training exercise
Other: Aerobic training exercise — randomized complete crossover for acute aerobic exercise training exercise session
  Arms: aerobic training exercise

SUMMARY:
The purpose of this study is to determine the effect of age and fitness level on the physiological response to an acute bout of resistance or aerobic exercise.

DETAILED DESCRIPTION:
Young and middle-aged to older adults who are physically active or not physically active will participate in two moderate to vigorous intensity exercise bouts: aerobic exercise and resistance training exercise. Blood will be collected to assess immune function and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* "Young" Adults: ages 18-30
* "Older" Adults: ages 55-75 and if a female postmenopausal
* Participants classified as "trained" must participate in at least 30 minutes of moderate to vigorous intensity cardiovascular activity at least 3 days per week and engage in resistance training for all of the major muscle groups approximately 2 days / week. They must have upheld this activity for the past 3 months
* Participants classified as "untrained" must be participating in less than 30 minutes of moderate to vigorous intensity cardiovascular activity and less than 2 days of resistance training per week for at least the last 3 months.

Exclusion Criteria:

* Have any contraindications to moderate to vigorous exercise
* Range of motion restrictions that would prevent them from participating in aerobic or resistance training with proper form (they must be ambulatory)
* aking medications (prescription or over the counter) known to influence immune function, including daily NSAID's, beta blockers, statins, bisphosphonates, or steroids.
* Have known cardiovascular, respiratory, metabolic, or renal disease, with the exception of controlled hypertension (as defined by resting BP below 140/90) and/or controlled asthma (self-reported).
* Be pregnant
* Be unable to complete all visits (i.e. must not be planning to leave the Houston area long-term before concluding their participation in the study which will span several weeks)
* Fall outside of a BMI range of (18.5 - 30)
* Consume alcohol or recreational drugs for 24h prior to visits
* Older women cannot be pre-menopausal (must have not had a menses for at least 12 months)
* Unable to speak or read English
* Participants must not have scheduling conflicts that would prevent them from reporting to the laboratory of integrated physiology 4 times over the course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Monocyte subset and function | Pre-resistance training (RT) exercise, change from pre-RT exercise to immediately post-RT exercise, change from pre-RT exercise to 1hr post-RT exercise, change from immediately post-RT exercise to 1hr post-RT exercise
  Flow cytometry to classify monocyte subsets and in vitro LPS stimulation to assess monocyte function
Monocyte subset and function | Pre-aerobic training (AT) exercise, change from pre-AT exercise to immediately post-AT exercise, change from pre-AT exercise to 1hr post-AT exercise, change from immediately post-AT exercise to 1hr post-AT exercise
  Flow cytometry to classify monocyte subsets and in vitro LPS stimulation to assess monocyte function
Monocyte subset and function | compare pre-RT to pre-AT
  Flow cytometry to classify monocyte subsets and in vitro LPS stimulation to assess monocyte function
Monocyte subset and function | compare immediately post-RT to immediately post-AT
  Flow cytometry to classify monocyte subsets and in vitro LPS stimulation to assess monocyte function
Monocyte subset and function | compare 1hr post-RT to 1hr post-AT
  Flow cytometry to classify monocyte subsets and in vitro LPS stimulation to assess monocyte function
NK cell function | Pre-resistance training (RT) exercise, change from pre-RT exercise to immediately post-RT exercise, change from pre-RT exercise to 1hr post-RT exercise, change from immediately post-RT exercise to 1hr post-RT exercise
  Flow cytometry to identify NK cells and in vitro activity to assess NK activity
NK cell function | Pre-aerobic training (AT) exercise, change from pre-AT exercise to immediately post-AT exercise, change from pre-AT exercise to 1hr post-AT exercise, change from immediately post-AT exercise to 1hr post-AT exercise
  Flow cytometry to identify NK cells and in vitro activity to assess NK activity
NK cell function | compare pre-RT to pre-AT
  Flow cytometry to identify NK cells and in vitro activity to assess NK activity
NK cell function | compare immediately post-RT to immediately post-AT
  Flow cytometry to identify NK cells and in vitro activity to assess NK activity
NK cell function | compare 1hr post-RT to 1hr post-AT
  Flow cytometry to identify NK cells and in vitro activity to assess NK activity
Circulating relative and absolute counts of T cell subsets | Pre-resistance training (RT) exercise, change from pre-RT exercise to immediately post-RT exercise, change from pre-RT exercise to 1hr post-RT exercise, change from immediately post-RT exercise to 1hr post-RT exercise
  Flow cytometry to identify T cell subsets
Circulating relative and absolute counts of T cell subsets | Pre-aerobic training (AT) exercise, change from pre-AT exercise to immediately post-AT exercise, change from pre-AT exercise to 1hr post-AT exercise, change from immediately post-AT exercise to 1hr post-AT exercise
  Flow cytometry to identify T cell subsets
Circulating relative and absolute counts of T cell subsets | compare pre-RT to pre-AT
  Flow cytometry to identify T cell subsets
Circulating relative and absolute counts of T cell subsets | compare immediately post-RT to immediately post-AT
  Flow cytometry to identify T cell subsets
Circulating relative and absolute counts of T cell subsets | compare 1hr post-RT to 1hr post-AT
  Flow cytometry to identify T cell subsets

SECONDARY OUTCOMES:
Serum cortisol | Pre-resistance training (RT) exercise, change from pre-RT exercise to immediately post-RT exercise, change from pre-RT exercise to 1hr post-RT exercise, change from immediately post-RT exercise to 1hr post-RT exercise
  ELISA to measure circulating cortisol (serum)
Serum cortisol | Pre-aerobic training (AT) exercise, change from pre-AT exercise to immediately post-AT exercise, change from pre-AT exercise to 1hr post-AT exercise, change from immediately post-AT exercise to 1hr post-AT exercise
  ELISA to measure circulating cortisol (serum)
Serum cortisol | compare pre-RT to pre-AT
  ELISA to measure circulating cortisol (serum)
Serum cortisol | compare immediately post-RT to immediately post-AT
  ELISA to measure circulating cortisol (serum)
Serum cortisol | compare 1hr post-RT to 1hr post-AT
  ELISA to measure circulating cortisol (serum)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Markofski, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are considering making available IDP to others upon request, but would have to get an IRB change because that is not in our protocol

REFERENCES:
- [Derived] Graff RM, Jennings K, LaVoy ECP, Warren VE, Macdonald BW, Park Y, Markofski MM. T-cell counts in response to acute cardiorespiratory or resistance exercise in physically active or physically inactive older adults: a randomized crossover study. J Appl Physiol (1985). 2022 Jul 1;133(1):119-129. doi: 10.1152/japplphysiol.00301.2021. Epub 2022 May 26. PMID 35616304